CLINICAL TRIAL: NCT05446311
Title: Naldebain® Extended-release Injection After Cesarean Section in Pain Management: a Prospective Observational Study
Brief Title: Naldebain® Extended-release Injection After Cesarean Section in Pain Management
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Chi-Kang Lin, Director, Tri-Service General Hospital
Other Study IDs: TSGH-OBS-111-01
Record Dates: First submitted 2022-06-30; First posted 2022-07-06 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: Post Operative Pain; Caesarean Section; Analgesia
Keywords: Dinalbuphine Sebacate; NALDEBAIN; Extended-release analgesics
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Breast milk
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DS group: Subjects going to receive dinalbuphine sebacate for post-cesarean section pain.
  Interventions: Drug: Dinalbuphine sebacate

INTERVENTIONS:
Drug: Dinalbuphine sebacate — After giving the birth, subjects are intramuscularly injected with a single dose of 150 mg of dinalbuphine sebacate (DS). DS is a prodrug of nalbuphine. After injeciton, DS are released to blood stream and hydrolyzed immediately. The onset of action is 12 to 24 hours and the analgesic effect can last about 5 to 7 days.
  Other Names: NALDEBAIN

SUMMARY:
Cesarean section is one of the surgeries most commonly leading to postoperative severe acute pain. It was reported that the mean worst pain intensity reached to 6.14 one day after cesarean section in Germany. Inadequate pain management may result in the cardiorespiratory complications, late recovery, and postoperative chronic pain. According to a series of pain management article published in the Lancent in 2019, the incidence of post-cesarean section chronic pain was 55%, including 12% of severe chronic pain. Extended-release dinalbuphine sebacate, a prodrug of nalbuphine, is a novel analgesic developed in Taiwan and the indication is moderate to severe postoperative pain. After intramuscular injected, dinalbuphine sebacate will be released to blood stream and immediately hydrolyzed. In Taiwan, dinalbuphine sebacate has been used for alleviating pain after several types of surgeries, such as colorectal surgery, orthopaedics, gynecology and obstetrics. However, few post-marketing studies investigated the efficacy and safety of dinalbuphine sebacate.

DETAILED DESCRIPTION:
This is an observational, prospective, single arm study. This study is aimed to investigate the efficacy and safety of dinalbuphine sebacate in subjects undergoing cesarean section. Written informed consent are obtained before subjects participate in the study. Eligible subjects will be visited twice daily during stay in hospital. Pain intensity, consumption of analgesics, adverse reaction, and the residues of dinalbuphine sebacate and nalbuphine in milk will all be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Female aged 20 to 45 years.
2. Going to have cesarean section and use dinalbuphine sebacate to alleviate postoperative pain.
3. Cesarean section scheduled between the 34th and 41st week of gestation.
4. ASA I or II.
5. Willing to comply with study protocol and give written informed consent.

Exclusion Criteria:

1. With contraindication to opioids.
2. Chronic use or abuse of opioids.
3. Underlying disease which contribute to abnormal lactation, such as mastitis.
4. Diagnosed with gestational diabetes mellitus and administration of insulin is required.
5. Diagnosed with pre-eclampsia or eclampsia.
6. Unsuitable for participation judged by investigator.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Subjects going to undergo cesarean section
Study Population: Subjects going to have cesarean section in Tri-Service General Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-07-15 (Estimated); Primary Completion 2022-12-20 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of complication | Within 5 days after injection of dinalbuphine sebacate
  Analgesic-related complication occurring in the period of hospital stay will be recorded, such as dizziness, nausea, vomiting, and injection site reaction.

SECONDARY OUTCOMES:
Post-cesarean section pain intensity | Within 5 days after delivery
  Pain intensity is assessed by numerical rating scale (NRS) twice daily during stay
Consumption of analgesics | Within 5 days after delivery
  Analgesics consumed during stay of hospital are recorded.
Concentration of nalbuphine in breast milk | Within 5 days after delivery
  Dinalbuphine sebacate is a prodrug of nalbuphine. After intramuscular injection, dinalbuphine sebacate are slowly released to blood stream and immediately hydrolyzed. The breast milk is collected twice daily within 5 days after cesarean section, and tested by HPLC.
Concentration of dinalbuphine sebacate in breast milk | Within 5 days after delivery
  Dinalbuphine sebacate is a prodrug of nalbuphine. After intramuscular injection, dinalbuphine sebacate are slowly released to blood stream and immediately hydrolyzed. The breast milk is collected twice daily within 5 days after cesarean section, and tested by HPLC.

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Kang Lin, MD, Principal Investigator — Tri-Service General Hospital